CLINICAL TRIAL: NCT05480397
Title: TRANSCUTANEOUS ELECTRICAL NERVE STIMULATION VERSUS DISTRACTIVE TECHNIQUES ON ARTERIOVENOUS FISTULA PUNCTURE PAIN IN HEMODIALYSIS PATIENTS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Gamal Abdelmohsen Abdelhakim Hassan, physical therapist, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P.T.REC/012/003723
Record Dates: First submitted 2022-07-27; First posted 2022-07-29 (Actual); Last update posted 2022-07-29 (Actual); Status verified 2022-07

CONDITIONS: TENS, Distractive Techniques, Arteriovenous Fistula, Puncture Pain, Hemodialysis
MeSH Terms: conditions — Arteriovenous Fistula | interventions — Transcutaneous Electric Nerve Stimulation; Cryotherapy

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- • Group (1) will receive (TENS , cryotherapy and conventional physical therapy program). (Experimental)
  Interventions: Other: TENS, Distractive techniques, cryotherapy
- •Group (2) receive (distractive techniques , cryotherapy and conventional physical therapy) (Experimental)
  Interventions: Other: TENS, Distractive techniques, cryotherapy
- • Group (3) will receive (cryotherapy and conventional physical therapy program). (Experimental)
  Interventions: Other: TENS, Distractive techniques, cryotherapy

INTERVENTIONS:
Other: TENS, Distractive techniques, cryotherapy — Group (1): Will receive (TENS , cryotherapy and conventional physical therapy ) Massage with ice was done by the researcher over the AVF puncture site . After that, the TENS electrodes will be applied by the researcher 6 centimeters apart closely up and down the skin area for insertion of the needle.
  * Group (2): Will receive (Distraction techniques ,cryotherapy and conventional physical therapy ) Initially five minutes before starting hemodialysis, Distraction techniques will be applied. Natural and eye-catching images were broadcasted through a video display device on a laptop monitor in a manner that was easy for the older patient to watch while they were lying on the bed. Massage with ice was done by the researcher over the AVF puncture site
  * Group (3): Will receive (cryotherapy and conventional physical therapy )

SUMMARY:
Statement of the problem:

This study will be conducted to answer the following question:

Is there a difference in the efficacy of TENS and distractive techniques when combined with cryotherapy in managing pain due to arteriovenous fistula puncture and improving quality of life in hemodialysis patients ?

Null Hypotheses:

1. TENS has no statistically significant effect on pain management and quality of life in hemodialysis patients undergoing arteriovenous fistula puncture.
2. Distractive techniques have no statistically significant effect on pain management and quality of life in hemodialysis patients undergoing arteriovenous fistula puncture.
3. There is no statistically significant difference between TENS and distractive techniques in managing pain and improving quality of life in hemodialysis patients undergoing arteriovenous fistula puncture.

DETAILED DESCRIPTION:
Subjects' Selection:

The patients will be randomly assigned to 3 groups;

* Group (1) will receive (TENS , cryotherapy and conventional physical therapy program).
* Group (2) will receive (distractive techniques , cryotherapy and conventional physical therapy program).
* Group (3) will receive (cryotherapy and conventional physical therapy program). Patients will be assessed for quality of life before and after treatment and will receive 3 sessions per week consisted of TENS, distractive techniques , Cryotherapy and conventional physical therapy program during AVF Puncture during dialysis for 4 weeks.

  1-Inclusion criteria:
  1. Patient age will range from 20 - 60 years who have chronic renal failure from males and females.
  2. At least one year passed from the installation of AVF and hemodialysis.
  3. Patients are undergoing hemodialysis three sessions per week and each session lasting for 4 hours.
  4. Having no traces of skin abnormalities or analgesia in vessels access point.

  2-Exclusion Criteria:

The following were considered exclusion criteria:

1. Unwillingness to continue with the study.
2. Unsuccessful AVF cannulation at the first try.
3. Patients having radiation injuries, peripheral vascular diseases, Raynauld's disease, connective tissue disorders, diabetic neuropathy, unconsciousness or disorientation.
4. Presence of infection and obstruction of fistula based on the nurse's inspection.
5. The presence of auditory and visual disturbances.
6. history of verbal disturbances; no addiction or drug dependence to pain medications; no history of mental health diseases; being conscious, having not taken painkillers, narcotics or sedatives at least six hours before hemodialysis.
7. Having traces of severe pain in other parts.
8. Having pacemakers. The patients will be randomly assigned to 3 groups; Group(1) will receive TENS , cryotherapy and conventional physical therapy program, Group(2) will receive distractive techniques , cryotherapy and conventional physical therapy program and Group(3) will receive cryotherapy and conventional physical therapy program.

All groups will be assessed for quality of life using Kidney Disease Quality of Life Short Form Scale (KDQOL-SF) before and after treatment.

ELIGIBILITY:
Inclusion Criteria:

* 1-Inclusion criteria:

  1. Patient age will range from 20 - 60 years who have chronic renal failure from males and females.
  2. At least one year passed from the installation of AVF and hemodialysis.
  3. Patients are undergoing hemodialysis three sessions per week and each session lasting for 4 hours.
  4. Having no traces of skin abnormalities or analgesia in vessels access point.

Exclusion Criteria:

* 2-Exclusion Criteria:

The following were considered exclusion criteria:

1. Unwillingness to continue with the study.
2. Unsuccessful AVF cannulation at the first try.
3. Patients having radiation injuries, peripheral vascular diseases, Raynauld's disease, connective tissue disorders, diabetic neuropathy, unconsciousness or disorientation.
4. Presence of infection and obstruction of fistula based on the nurse's inspection.
5. The presence of auditory and visual disturbances.
6. history of verbal disturbances; no addiction or drug dependence to pain medications; no history of mental health diseases; being conscious, having not taken painkillers, narcotics or sedatives at least six hours before hemodialysis.
7. Having traces of severe pain in other parts.
8. Having pacemakers

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 45 (Estimated)
Dates: Start 2022-06-15 (Actual); Primary Completion 2022-09 (Estimated); Study Completion 2022-10 (Estimated)

PRIMARY OUTCOMES:
The KDQOL-36, Numerical Rating Scale for pain measurement | one hour for each participant
  1. Numerical Rating Scale of Pain Severity is numbered between 0 and 10 indicating positive and negative pain statements, respectively. Accordingly, the rating of this scale was 0 (lack of pain), 1-3 (low pain), 4-6 (moderate pain), 7-9 (severe pain), and 10 (very severe pain). The Cronbach's alpha coefficient for this tool was reported as 0.95 and its reliability score using the intra-class correlation coefficient was 0.92 (Mirtajadini et al., 2016).
  2. The KDQOL-36:
  It is a 36-item health-related quality of life instrument adapted from the original 134-item KDQOL, an instrument principally developed to measure quality of life of dialysis patients [25].

CONTACTS AND LOCATIONS:
Locations (1):
- Hemodialysis unit, General Ashmoon Hospital, Ashmoon, Menofia, Menofia, Egypt